CLINICAL TRIAL: NCT05310305
Title: Combination of Immune Checkpoint Inhibitors PD-1 Monoclonal Antibody and Radiotherapy for Recurrent, Metastatic and Persistent Advanced Cervical Cancer: A Retrospective Cohort Study
Brief Title: PD-1 Antibody and Radiotherapy for Recurrent Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: IMURADIO1
Record Dates: First submitted 2022-03-26; First posted 2022-04-04 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Immune Checkpoint Inhibitors; Anti-programmed Death-1 Antibody; Radiotherapy; Recurrent Cervical Carcinoma; Metastatic Cervical Carcinoma; Persistent Advanced Cervical Carcinoma; Objective Remission Rate; Progression-free Survival; Overall Survival; Severe Adverse Events
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Radiotherapy for targeted lesions and PD-1 antibody — Radiotherapy for targeted lesions in all enrolled participants, with concurrent PD-1 antibody. Patients may or may not accept subsequent PD-1 as maintenance therapy.

SUMMARY:
This study is to investigate retrospectively the effects of combination of immune checkpoint inhibitors anti-programmed death-1 antibody (PD-1 antibody) and radiotherapy for recurrent, metastatic and persistent advanced cervical carcinomas. Patients may or may not accept PD-1 antibody as maintenance therapy. Patients are followed up and the survival outcomes are evaluated. The primary endpoint are objective remission rate. The secondary endpoints are progression-free survival, overall survival and severe adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Confirmed of recurrent, metastatic, and persistent advanced cervical cancer
* Confirmed of subtypes of cervical squamous carcinoma, adenocarcinoma and adenosquamous carcinoma
* Accepting radiotherapy with concurrent anti PD-1 therapy
* With detailed follow-up outcomes

Exclusion Criteria:

- Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent, metastatic and persistent advanced cervical carcinomas
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-03-26 (Actual); Primary Completion 2022-09-26 (Estimated); Study Completion 2023-03-26 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate | One year
  Objective remission rate in one month after the end of radiotherapy

SECONDARY OUTCOMES:
Progression-free survival | One year
  Progression-free survival after the end of radiotherapy
Overall survival | One year
  Overall survival after the end of radiotherapy
Severe adverse events | Two years
  Severe adverse events during the radiotherapy and the follow-up stage

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China